CLINICAL TRIAL: NCT03833752
Title: Randomized Controlled Study To Evaluate The Outcomes Between Rigid And Flexible Cystoscopy In Men With Lower Urinary Tract Symptoms Undergoing Diagnostic Cystoscopy
Brief Title: Flexible V/S Rigid Cystoscopy In Men With Urinary Tract Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maulana Azad Medical College (Other)
Responsible Party: Principal Investigator, Dr. Gaurish Sawant, resident doctor, Maulana Azad Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: F.No./11IEC/MAMC/2016/113
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: rigid cystoscopy; flexible cystosocpy; UTI; BPH
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible Cystoscopy (Experimental): Diagnostic flexible cystoscopy for the patients in this arm
  Interventions: Diagnostic Test: Diagnostic Flexible Cystosocpy
- Rigid Cystoscopy (Active Comparator): Diagnostic rigid cystoscopy is done for the patients in this arm
  Interventions: Diagnostic Test: Diagnostic Rigid Cystoscopy

INTERVENTIONS:
Diagnostic Test: Diagnostic Flexible Cystosocpy — Endoscopic Visualization of the Lower Urinary tract using either a flexible cystoscope for the purpose of aiding the establishment of a Urological Diagnosis.
  Arms: Flexible Cystoscopy
Diagnostic Test: Diagnostic Rigid Cystoscopy — Endoscopic Visualization of the Lower Urinary tract using either a rigid cystoscope for the purpose of aiding the establishment of a Urological Diagnosis.
  Arms: Rigid Cystoscopy

SUMMARY:
The objective of this study is to perform a randomized study, comparing the outcomes of the above two types of cystoscopy in terms of discomfort experienced by the patient, while undergoing the procedure.

DETAILED DESCRIPTION:
Cystoscopy is a commonly performed routine outpatient procedure and an essential diagnostic tool in urology.Compared with flexible endoscopes, rigid instruments offer better image quality, a wider lumen of the working channel, improved irrigant flow and superior handiness. However, flexible cystoscopes provide more options for patient positioning, enable smooth passage over an elevated bladder neck or median lobe, facilitate full inspection of the bladder because of their movable tip and, what is most important is it significantly improve patient comfort(patient can be positioned in any comfortable position).

ELIGIBILITY:
Inclusion Criteria:

* patients with lower urinary tract symptoms

Exclusion Criteria:

* patients with Suprapubic catheter
* History of radical prostatectomy or cystoprostatectomy
* Clinical evidence of urethral stricture, prostatitis
* Patients with bacterial growth on urine culture

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
Post Procedure Discomfort | periprocedure
  Discomfort experienced immediately post procedure by the patient defined as a Visual Analogue Scale score of more than 3 (range is from 1 to 10)
Duration of Procedure | periprocedure
  time taken to complete the entire test in minutes starting from insertion of the cystoscope through the urethral meatus, visualising the entire bladder and urethra , till the removal of the scope after making the observations.

CONTACTS AND LOCATIONS:
Overall Officials: PAWAN LAL, MS,DNB,DA, Study Director — Professor, Department of Surgery
Locations (1):
- Maulana Aazad Medical College, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared to all researchers who produce the query for it.
Supporting Information: Study Protocol, SAP, ICF, CSR